CLINICAL TRIAL: NCT02192203
Title: Safety Study to Investigate the Skin Sensitization Potential of MFC51123
Brief Title: A Safety Study to Investigate the Skin Sensitization Potential of MFC51123
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 202186; RH02169 (Other: GSK)
Record Dates: First submitted 2014-05-15; First posted 2014-07-16 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diclofenac + Menthol Gel (Experimental): 1% diclofenac, 3% menthol
  Interventions: Drug: Diclofenac + Menthol Gel
- Diclofenac Only Gel (Active Comparator): 1% diclofenac, 0.09% menthol
  Interventions: Drug: Diclofenac Only Gel
- Menthol Only Gel (Active Comparator): 3% menthol
  Interventions: Drug: Menthol Only Gel
- Placebo Only Gel (Placebo Comparator): 0.09% menthol
  Interventions: Drug: Placebo Only Gel

INTERVENTIONS:
Drug: Diclofenac + Menthol Gel — 1% diclofenac, 3% menthol
  Arms: Diclofenac + Menthol Gel
Drug: Diclofenac Only Gel — 1% diclofenac, 0.09% menthol
  Arms: Diclofenac Only Gel
Drug: Menthol Only Gel — 3% menthol
  Arms: Menthol Only Gel
Drug: Placebo Only Gel — 0.09% menthol
  Arms: Placebo Only Gel

SUMMARY:
This research study is being carried out to determine the possibility that a new medication causes allergic reactions. This new medication contains two active ingredients (diclofenac and menthol) together in a gel and is being developed to treat mild to moderate pain and inflammation, such as acute sport injuries, and sprains and strains. Approximately 240 participants will have the medication (gel) applied to the skin on a small area of the upper back for approximately 48-hour or 72-hour periods over the course of six weeks. Participation in this research study is voluntary, requiring participants to visit the study clinic on 17 occasions for about 45 minutes each visit. During the visits, doctors or trained staff members will examine the amount of redness, swelling, and other signs of irritation (if any) of the skin where the medication (gel) was applied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women participants with 18 years of age or older.

Exclusion Criteria:

* Participants with a history of hypersensitivity, allergy with the use of NSAIDs or menthol or currently receiving systemic or topical NSAIDs within 3 days of visit 1.
* Participants having psoriasis and/or active atopic dermatitis/eczema, and skin infected.
* Lesions, burn or wound in the application site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2014-07-15 (Actual); Study Completion 2014-07-15 (Actual)

PRIMARY OUTCOMES:
Skin irritation | At least 23 days but not more than 30 days for induction and challenge phases combined
  During the Induction Phase, the test article and three controls will be applied to adjacent treatment sites on the infrascapular area of the back for nine 48-hour patch applications. Evaluation of dermal reactions at the application sites will be conducted clinically using a visual scale that rates the degree of erythema, edema, and other signs of cutaneous irritation at nine intervals spaced approximately 48-72 hours apart. Following the Induction Phase participants will return to the clinic to begin the Challenge Phase after 12 to 14- day rest phase. The Challenge Phase will consist of one 48-hour patch application to a naive site on the opposite side of the back. Evaluations of dermal reactions at the application sites will be conducted clinically during the Challenge Phase using the same visual scale at 30 minutes, 24 hours, 48 hours, and 72 hours after removal of the challenge patch.

SECONDARY OUTCOMES:
Effects on Superficial Layers of the Skin | At least 23 days but not more than 30 days for induction and challenge phases combined
  The responses will be assessed using symbol (A-H) and grade (0 -3) scale for each of the four test products: A 0 Slight glazed appearance; C 1 Marked glazing; E 2 Glazing with peeling and cracking; F 3 Glazing with fissures; G 3 Film of dried serous exudate covering all or portion of the patch; H 3 Small petechial erosions and/or scabs
Response notation | At least 23 days but not more than 30 days for induction and challenge phases combined
  Notations will be made in place of a score to designate particular circumstances preventing the assignment of a score or in addition to a score to identify damage to the epidermis and/or spreading of a reaction beyond the patch site.S: Spreading of reaction beyond patch study site (i.e., reaction where study material was not in contact with the skin); B: Burning or stinging sensation; P: Papular response >50%; Pv: Papulovesicular response >50%; D: Damage to epidermis: oozing, crusting and/or superficial erosions; I; Itching; X: absent Subject absent; PD: Patch dislodged; NA Not applied; NP: Not patched (due to reaction achieved); N9G: No ninth grading

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- TKL Research Inc, Paramus, New Jersey, United States

REFERENCES:
- See also: Results for the study 202186 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/202186?search=study&search_terms=202186#rs